CLINICAL TRIAL: NCT02488226
Title: Gaze Modification Strategies for Toddlers With Autism Spectrum Disorder
Acronym: ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Frederick Shic, Assistant Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1306012246
Record Dates: First submitted 2015-06-24; First posted 2015-07-02 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gaze Contingent (Experimental): Participants will view social videos using Gaze-contingent eye-tracking technology . If the participants looking patterns deviate from a normative pattern, they will be redirected to the normative point of regard using gaze-contingent cues.
  Interventions: Other: Gaze-contingent eye-tracking technology
- Control Condition (No Intervention): Participants will view unaltered social videos which do not change based on where the participant is looking.

INTERVENTIONS:
Other: Gaze-contingent eye-tracking technology — When participants look away from a prototypical or expected norm, their gaze patterns are redirected to those prototypical locations.
  Arms: Gaze Contingent

SUMMARY:
This project seeks to understand how the gaze behavior of infants and children with or at high risk for autism spectrum disorder (ASD) may be manipulated in the contexts of dynamic social and non-social scenes. The study explores not only the methods which may be most effective in aligning and teaching normative patterns of scene exploration, but also seeks to establish what behavioral characteristics may be most predictive of atypical scanning and atypical learning.

DETAILED DESCRIPTION:
This study initiates a highly novel line of research which uses adaptive, gaze-contingent, eye-tracking technology to help infants and children with or at high risk for ASD learn to direct their attention to people and their actions in a more typical fashion. This study will begin with a Normative Collection phase, and will conclude with a Gaze-Shaping phase. In the Normative Collection phase, the investigators will examine the gaze behavior of a group of typically developing infants and children with typical development (TD), in order to establish a normative gaze pattern. In the Gaze-Shaping phase, within the same videos shown in the Normative Collection phase, the investigators will highlight selectively targeted people, objects, and activities, in an attempt to shape participants' viewing patterns to match the normative gaze pattern.

Manual coding of live-action interaction probes will provide an additional evaluative measure, allowing the investigators to track real-world (live-action) correlates alongside video-eye-tracking behaviors. In addition, live-action probes may allow the investigators to check for generalization to live interaction with another person (as opposed to gaze behavior when watching videos). In live-action probes, one or two clinical research staff member(s) will interact with each participant (or with each other in front of the participant), in a manner analogous to the actions performed in the training videos.

Please note: The original estimated enrollment as specified to and funded by NIH was 98 participants, but was incorrectly listed on ClinicalTrials.gov as 220 participants reflecting maximal recruitment in this and other ongoing studies.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 60 months
* Fulfill criteria for autistic disorder or PDD-NOS (Pervasive Developmental Disorder- Not Otherwise Specified) on the Autism Diagnostic Observation Schedule - Module 1
* A diagnosis of autism or PDD-NOS by experienced clinicians

Exclusion Criteria:

* Gestational age below 32 weeks
* Suspected or diagnosed hearing loss or visual impairment
* History of head trauma with loss of consciousness
* Non-febrile seizure disorders
* Diagnosed neurological abnormality significantly impacting on visual or auditory acuity.

Ages: 18 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Gaze behavior during eye tracking tasks measured by standard eye-tracking analysis protocols | 1-7 days
  Outcome measures for eye-tracking will include the Percentage of Time Spent Looking at Face, Body, and Background regions for stimuli involving people, and Percentage of Time Spent Looking at Activity, People, and Background regions. Percentage of time spent looking at the video (i.e. overall attention less motion, blinks, and inattention) will be calculated. Additional variables specific to the training sessions' adaptive cue condition will include the number of times the stimuli is adapted to redirect attention to locations consistent with the typical viewing pattern) and the amount of time spent in redirection. These will all be assessed by standard eye-tracking analysis protocols.

SECONDARY OUTCOMES:
Behavior during real-world interactions measured by coding of video recordings | 1-7 days
  Outcome measures include attention to social interactions and responses bids for engagement in social attention during a live experimental session, as measured by coding of video recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Shic, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States